CLINICAL TRIAL: NCT04573465
Title: Pilot Evaluation of Peer-support Coaching to Increase Adherence to Online Self-help for College Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Michael Levin, Associate Professor, Utah State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11308
Record Dates: First submitted 2020-09-27; First posted 2020-10-05 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Treatment Adherence
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned with equal likelihood to receive the online intervention with coaching delivered through weekly phone calls, the online intervention with coaching delivered through weekly text messages, or the online intervention with no coaching.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phone Coaching Condition (Experimental): Participants will receive weekly, 10-15 minute phone coaching from a trained peer-support coach throughout the 10 weeks that they use ACT Guide, an online program for general mental health. Coaches will adhere to an ACT-based protocol that includes reinforcing adherence, identifying and problem solving non-adherence, strengthening and generalizing ACT skills, and using ACT skills to increase commitment to ongoing program adherence.
  Interventions: Behavioral: Phone Coaching; Behavioral: ACT Guide
- Text Message Coaching Condition (Experimental): Participants assigned to the text messaging condition will receive weekly text messages from their peer-support coach throughout the 10 weeks that they use ACT Guide, an online program for general mental health. These text messages will reflect content delivered in the phone coaching group, but through a briefer protocol that accounts for the abbreviated, asynchronous nature of texting. Text messages will similarly focus on reinforcing adherence, problem solving non-adherence, strengthening ACT skills, and using ACT to increase program adherence. However, these areas will be covered in short messages and with limited exchanges between participants and coaches due to the asynchronous nature of texting.
  Interventions: Behavioral: Text Message Coaching; Behavioral: ACT Guide
- No Coaching Condition (Active Comparator): Participants will be asked to use ACT Guide, an online program for general mental health, over the course of 10 weeks while receiving no coaching.
  Interventions: Behavioral: ACT Guide

INTERVENTIONS:
Behavioral: Phone Coaching — Participants receiving phone coaching receive one 10-15 minute phone call each week from their randomly assigned peer-support coach. During coaching calls, the peer-support coach will discuss ACT Guide usage with the participant (e.g., asking how many modules the participant completed, asking what the participant liked/disliked about the modules, etc.).
  Arms: Phone Coaching Condition
Behavioral: Text Message Coaching — Participants receiving text message coaching receive text messages on a weekly basis from their randomly assigned peer-support coach. Text messages from the peer-support coach will discuss ACT Guide usage with the participant (e.g., asking how many modules the participant completed).
  Arms: Text Message Coaching Condition
Behavioral: ACT Guide — ACT Guide is an online self-help program based on acceptance and commitment therapy (ACT), targeting acceptance, mindfulness, and values-based processes. It is intended to be used for 20 to 40 minutes at time, a few times a week. While using ACT Guide, participants will read about concepts relevant to ACT and engage in guided experiential exercises, with additional exercises being assigned to be completed in between sessions as homework.

SUMMARY:
This study aims to test if coaching can improve program adherence to an online mental health program in college students if delivered by undergraduate peers. Participants will be randomly assigned to either receive phone coaching, text message coaching, or no coaching. It is hypothesized that participants who receive phone coaching will exhibit greater adherence to the provided online mental health program than participants who receive text message coaching or no coaching.

DETAILED DESCRIPTION:
The purpose of this study is to test the feasibility and effectiveness of an innovative peer support coaching model for college students. The primary aim of the coaching model is to increase participants' adherence to ACT Guide, an online mental health program. To test the effects of peer-support coaching on ACT Guide adherence rates and outcomes, the investigators will conduct a randomized controlled trial with three conditions (peer-support phone coaching, peer-support text message coaching, and a no support control group) using a sample of 300 Utah State University undergraduate students. Individuals who indicate interest in participating will complete an automated online workflow through Qualtrics which will include informed consent, baseline assessment, ACT Guide registration, and randomization into one of the three conditions. Participants will then gain access to a research version of ACT Guide, either with no additional support, with concurrent peer-support coaching, or with concurrent peer-support text messaging based on their randomly assigned condition. Coaching will take place over 10 weeks, with the post assessment being administered 10 weeks after baseline assessment. The investigators hypothesize that participants will adhere to coaching (80% completing ≥ 6 coaching calls; 80% responding to texts > 6 weeks), be satisfied with coaching (M = 5 "agree" on a 6-point self-reported coaching satisfaction scale), and that coaching fidelity will be maintained (80% of audited coaching calls/texts meeting criteria for fidelity). The investigators also hypothesize that participants who receive peer-support phone coaching will complete more ACT Guide modules and will report greater improvements in mental health relative to both the text messaging and no support conditions, and that the text messaging condition will perform greater in this regard than the no support condition.

ELIGIBILITY:
Inclusion Criteria:

* USU undergraduate student
* Fluent in English

Exclusion Criteria:

* Must have not used ACT Guide in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
ACT Guide Module Completion | Post-treatment (10 weeks after baseline)
  Number of modules completed within ACT Guide, out of a total of 12 modules. This is automatically recorded within the ACT Guide program, and is not self-reported.
Depression, Anxiety, and Stress Scale (DASS-21; Osman et al., 2012) | Post-treatment (10 weeks after baseline)
  A self-report measure for depression, anxiety, and stress . Items are rated on a 4-point Likert scale from 0 (did not apply to me at all) to 3 (applied to me most of the time), with a higher score indicating a worse outcome. Minimum total of 0 and maximum total of 63.

SECONDARY OUTCOMES:
Short Form of the Revised Vanderbilt Therapeutic Alliance Scale adapted for coaching (VTAS-R; Shelef & Diamond, 2008) | After completion of first contact with coach and post-treatment (10 weeks after baseline)
  A self-report measure for therapeutic alliance, with modified wording in order to adapt to a coaching context. Only administered to participants in either coaching condition. Items are rates on a 6-point Likert scale from 0 (not at all) to 5 (a great deal), with a higher score indicating a better outcome. Minimum total of 0 and maximum total of 25.
Mental Health Continuum Short Form (MHC-SF; Keyes, 2005) | Post-treatment (10 weeks after baseline)
  A self-report measure for positive mental health. Items are rated on a 6-point Likert scale from 1 (never) to 6 (every day), with a higher score indicating a better outcome. Minimum total of 14 and maximum total of 84.
The Acceptance and Action Questionnaire (AAQ-II; Bond et al., 2011) | Post-treatment (10 weeks after baseline)
  A self-report measure for psychological flexibility. Items are rated on a 7-point Likert scale from 1 (never true) to 7 (always true), with a higher score indicating a worse outcome. Minimum total of 7 and maximum total of 49.
Comprehensive assessment of Acceptance and Commitment Therapy processes (CompACT; Francis, Dawson, & Golijani-Moghaddam, 2016) | Post-treatment (10 weeks after baseline)
  A self-report measure for psychological flexibility. Items are rated on a 7-point Likert scale from 0 (strongly disagree) to 6 (strongly agree), with a higher score indicating a better outcome. Minimum total of 0 and maximum total of 138.
Client Satisfaction Questionnaire adapted to Internet-based interventions (CSQ-I; Boß et al., 2016) | Post-treatment (10 weeks after baseline)
  A self-report measure for program satisfaction. Items are rated on a 4-point Likert scale from 1 (does not apply to me) to 4 (does totally apply to me), with a higher score indicating a better outcome. Minimum total of 8 and a maximum total of 32.
Novel user experience item 1 | Post-treatment (10 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "Overall, I was motivated to use ACT Guide" This is a user experience item specific to this study.
Novel user experience item 2 | Post-treatment (10 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "I had the support I needed to use ACT Guide." This is a novel user experience item specific to this study.
Novel user experience item 3 | Post-treatment (10 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "I understood the concepts and skills presented in ACT Guide." This is a novel user experience item specific to this study.
Novel user experience item 4 | Post-treatment (10 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "I was able to apply skills I learned in ACT Guide to my personal struggles and daily life." This is a novel user experience item specific to this study.
Novel user experience item 5 | Post-treatment (10 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "I was able to identify and problem solve barriers to using ACT Guide." This is a novel user experience item specific to this study.
Novel user experience item 6 | Post-treatment (10 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "Many college students who struggle with mental health issues use self-help resources like ACT Guide for support." This is a novel user experience item specific to this study.
Novel user experience item 7 | Post-treatment (10 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "People would judge me negatively if they found out I was using ACT Guide." This is a novel user experience item specific to this study.
Novel user experience item 8 | Post-treatment (10 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "College students approve of the use of self-help resources like ACT Guide for addressing mental health issues." This is a novel user experience item specific to this study.
Novel coaching experience item 1 | Post-treatment (10 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "I would have preferred using ACT Guide without a coach." This is a novel coaching experience item specific to this study. Only administered to participants in either coaching condition.
Novel coaching experience item 2 | Post-treatment (10 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "ACT Guide would have been just as helpful to me without a coach." This is a novel user experience item specific to this study. Only administered to participants in either coaching condition.
Novel coaching experience item 3 | Post-treatment (10 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "I would have preferred to receive coaching from a mental health professional." This is a novel user experience item specific to this study. Only administered to participants in either coaching condition.
Novel coaching acceptability item 1 | Post-treatment (10 weeks after baseline)
  Participants will be asked to rate "Coaching through phone calls" on a scale from 1 (Unacceptable) to 5 (Strongly preferred). This is a novel coaching acceptability item specific to this study. Only administered to participants in either coaching condition.
Novel coaching acceptability item 2 | Post-treatment (10 weeks after baseline)
  Participants will be asked to rate "Coaching through text messaging" on a scale from 1 (Unacceptable) to 5 (Strongly preferred). This is a novel coaching acceptability item specific to this study. Only administered to participants in either coaching condition.
Novel coaching acceptability item 3 | Post-treatment (10 weeks after baseline)
  Participants will be asked to rate "Coaching through email" on a scale from 1 (Unacceptable) to 5 (Strongly preferred). This is a novel coaching acceptability item specific to this study. Only administered to participants in either coaching condition.
Novel coaching acceptability item 4 | Post-treatment (10 weeks after baseline)
  Participants will be asked to rate "Coaching through videoconferencing software" on a scale from 1 (Unacceptable) to 5 (Strongly preferred). This is a novel coaching acceptability item specific to this study. Only administered to participants in either coaching condition.
Novel coaching satisfaction item 1 | Post-treatment (10 weeks after baseline)
  Participants will be asked "What was helpful about the coaching process?" to gather qualitative feedback on their respective coaching intervention. Only administered to participants in either coaching condition.
Novel coaching satisfaction item 2 | Post-treatment (10 weeks after baseline)
  Participants will be asked "What was unhelpful about the coaching process?" to gather qualitative feedback on their respective coaching intervention. Only administered to participants in either coaching condition.
Novel coaching satisfaction item 3 | Post-treatment (10 weeks after baseline)
  Participants will be asked "How did having another USU undergraduate be your coach affect the coaching process?" to gather qualitative feedback on their respective coaching intervention. Only administered to participants in either coaching condition.
Novel coaching satisfaction item 4 | Post-treatment (10 weeks after baseline)
  Participants will be asked "How can the coaching process be improved in the future?" to gather qualitative feedback on their respective coaching intervention. Only administered to participants in either coaching condition.
Phone coaching adherence | Post-treatment (10 weeks after baseline)
  Number of coaching calls answered, out of a total of 10 calls. This is based on coaches call logs, and is not self-reported. Only applicable to participants in the phone coaching condition.
Text coaching adherence | Post-treatment (10 weeks after baseline)
  Number of initial coaching text messages responded to, out of a total of 10 initial text messages (one sent per week, not including text messages continuing a conversation stemming from an initial text message). This is based on coaches text message logs, and is not self-reported. Only applicable to participants in the text message coaching condition.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Levin, PhD, Principal Investigator — Utah State University
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boss L, Lehr D, Reis D, Vis C, Riper H, Berking M, Ebert DD. Reliability and Validity of Assessing User Satisfaction With Web-Based Health Interventions. J Med Internet Res. 2016 Aug 31;18(8):e234. doi: 10.2196/jmir.5952. PMID 27582341
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Francis A, Dawson D, Golijani-Moghaddam N. The development and validation of the Comprehensive assessment of Acceptance and Commitment Therapy processes (CompACT). Journal of Contextual Behavioral Science. 2016; 5(3): 134-145.
- [Background] Keyes CL. Mental illness and/or mental health? Investigating axioms of the complete state model of health. J Consult Clin Psychol. 2005 Jun;73(3):539-48. doi: 10.1037/0022-006X.73.3.539. PMID 15982151
- [Background] Osman A, Wong JL, Bagge CL, Freedenthal S, Gutierrez PM, Lozano G. The Depression Anxiety Stress Scales-21 (DASS-21): further examination of dimensions, scale reliability, and correlates. J Clin Psychol. 2012 Dec;68(12):1322-38. doi: 10.1002/jclp.21908. Epub 2012 Aug 28. PMID 22930477
- [Background] Levin ME, Krafft J, Hicks ET, Pierce B, Twohig MP. A randomized dismantling trial of the open and engaged components of acceptance and commitment therapy in an online intervention for distressed college students. Behav Res Ther. 2020 Mar;126:103557. doi: 10.1016/j.brat.2020.103557. Epub 2020 Jan 22. PMID 32014692
- [Background] Levin ME, Haeger JA, Pierce BG, Twohig MP. Web-Based Acceptance and Commitment Therapy for Mental Health Problems in College Students: A Randomized Controlled Trial. Behav Modif. 2017 Jan 1;41(1):141-162. doi: 10.1177/0145445516659645. Epub 2016 Jul 20. PMID 27440189
- [Background] Shelef K, Diamond GM. Short form of the revised Vanderbilt therapeutic alliance scale: development, reliability, and validity. Psychother Res. 2008 Jul;18(4):433-43. doi: 10.1080/10503300701810801. PMID 18815995
- [Background] Shim M, Mahaffey B, Bleidistel M, Gonzalez A. A scoping review of human-support factors in the context of Internet-based psychological interventions (IPIs) for depression and anxiety disorders. Clin Psychol Rev. 2017 Nov;57:129-140. doi: 10.1016/j.cpr.2017.09.003. Epub 2017 Sep 12. PMID 28934623